CLINICAL TRIAL: NCT03592602
Title: Evaluate the Impact of Arm Abduction and Adduction on the Intravascular Electrocardiograph During PICC Placement and the Tip Location Changes Related to it
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 26010105051802
Record Dates: First submitted 2018-07-01; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Catheterization, Peripheral; Catheterization, Central Venous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- arm movement (Experimental): Male or female patients, age ≥ 18, who meet the indication of PICC placement and be able to move the arm (abducted and adducted) with compliance will be studied.
  Interventions: Procedure: arm abduction and adduction

INTERVENTIONS:
Procedure: arm abduction and adduction — All PICC lines will be placed under the guidance of intravascular ECG. Before the PICC placement procedure, basal ECG will be examed. During the procedure, intravascular ECG data will be collected with the punctured arm adduction and abduction while the catheter advances to the cavoatrial junction. After the procedure, chest X-ray radiographs will be taken with arms 90° abducted and adducted (i.e., 0°abducted) in a supine position.

SUMMARY:
The purpose of the study is to evaluate the impact of arm abduction and adduction on the intravascular electrocardiograph during PICC placement and to find out how arm position influences the catheter tip location by taking postprocedural chest X-ray radiographs.

DETAILED DESCRIPTION:
PICC has been widely applied for therapeutic and nutritional use. In the routine procedure of PICC placement, for better exposure of the punctured vein and a wider aseptic area, the PICC set is investigated with the patient's arm abducted in a supine position. While in actual use of the PICC line, patients commonly prefer a more comfortable position with arm adducted. Considering the incorporation of the arm position when the catheter is placed and being used, the effectiveness and safety of the PICC line with the punctured arm adducted are of practical importance.

This study aims to evaluate the impact of arm abduction and adduction on the intravascular electrocardiograph (ECG) during ECG-guided PICC placement and to explore how arm movement (from abduction to adduction) makes an influence on the catheter tip position.

This study is expected to enroll 150 participants. All participants would undergo the procedure of ECG-guided PICC placement. ECG data will be recorded before the procedure (basal ECG) and during the procedure with the punctured arm abducted and adducted. After the procedure, participants will take a post chest X-ray confirmation with arms adducted and abducted in a supine position. The catheter tip position and influences of arm movements will be calculated by the distances from the catheter tip to the carina on radiographs.

ELIGIBILITY:
Inclusion Criteria:

* indication for PICC placement
* able to corporate with the operator during the procedure
* a recognizable P wave on basal ECG

Exclusion Criteria:

* bedside PICC placement
* Atrial fibrillation or other atrial arrhythmia's in which a P wave was not consistently present on ECG.
* with pacemaker
* unable to move to take post-procedural chest X-ray radiographs
* unable to move the punctured arm or can only move with limited angles due to anatomical abnormalities or personal/medical equipment or surgeries.
* catheter tip cannot be clearly visible on chest X-ray radiograph due to thoracic abnormalities or cardiothoracic surgeries.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-10-15 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
Changes of the intravenous ECG with the arm abducted and adducted during PICC placement. | Usually the procedure will take from 0-60 minutes.
  Comparing the shape and amplitude of the p wave with the arm abducted and adducted.

SECONDARY OUTCOMES:
Changes of the catheter tip position with the arm abducted and adducted. | Usually from 0-7 days after the procedure.
  Each patient will take two chest X-ray graphs with arms abducted and adducted respectively. Measuring distances from the catheter tip to the carina on radiographs.

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No